CLINICAL TRIAL: NCT05370222
Title: Adaptations of Exercise Energy Metabolism in Response to Simulated Weight Loss Versus Effective Weight Loss Induced by Diet in Healthy Normal Weight
Brief Title: Adaptations of Exercise Energy Metabolism in Response to Weight Loss in Healthy Normal Weight People
Acronym: NUTRILEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RBHP 2022 DUCLOS
Record Dates: First submitted 2022-05-02; First posted 2022-05-11 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Healthy; Weight Loss; Body Weight; Diet Habit; Healthy Nutrition
MeSH Terms: conditions — Weight Loss; Body Weight; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Behavioral: Dietary weight loss intervention

INTERVENTIONS:
Behavioral: Dietary weight loss intervention — Based on an energy assessment from the data collected at T0 (energy intake, physical activity level, and resting metabolism), individualized nutritional advice will be given during an interview in order to propose a dietary rebalancing and a light caloric restriction. Caloric restriction will be generated to decrease body weight by ≈ 0.5 to 1 kg per week, as advised in several publications. As for the dietary rebalancing, it will concern in particular the distribution of macronutrients and their nature (glycemic index, nature of lipids), the fibers intake, or the reduction of consumption of refined and/or energy-dense foods based on the ANSES Recommended Dietary Allowances and on the food consumption guidelines of the National Nutrition and Health Program.

SUMMARY:
More and more normal weight people are dieting in the general population. The NUTRILEX study aims to better understand the physiological adaptations in response to weight loss in healthy normal weight individuals.

After an inclusion visit to verify the eligibility criteria of the subjects, they will complete a "T0" control session. The subjects will then have to complete two phases. The first transversal phase consists of 4 randomized sessions with lunch ad libitum after a physical exercise: i) a control session (no exercise, CON); ii) an exercise session at initial body weight (BWT0); iii) an exercise session with a simulated weight loss of 3% performed on an anti-gravity treadmill (BW-3%) and; iv) an exercise session with a simulated weight loss of 6% performed on an anti-gravity treadmill (BW-6%).

During the second longitudinal phase, the participants will perform a dietary rebalancing and a slight caloric restriction (dietary intervention) in order to induce a weight loss of 6% of their initial body weight. Subjects will then perform an exercise session after losing 3% (T1) and then 6% (T2) of their initial body weight.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 and 24.9 kg/m²,
* Subjects abled to understand the information note and abled to sign the consent form,
* Subjects with stable body weight (variation < 3% of body weight) until at least 6 months,
* Subjects subjected to a social security plan.

Non-Criteria:

* Have achieved a minimal BMI < 18.5 or maximal BMI ≥ 25 kg/m² in adult life,
* Subjects with high levels of physical activity (> 5 h of exercise per week),
* Presence of comorbidities or medical conditions that may interfere with study data,
* Subjects undergoing energy restriction or physical activity weight loss program at the time of inclusion or within the past 6 months,
* Taking medication that may interfere with study results,
* Surgery within the last 3 months,
* Person under guardianship, curatorship, or safeguard of justice; or not subject to a social security plan,
* Pregnant or breastfeeding women,
* Refusal to sign the consent form,
* Person in a period of exclusion from another study,
* Regular consumption of tobacco or alcohol,
* Voluntary weight loss in the last 6 months,
* Present or past eating disorders.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2025-09-26 (Estimated); Study Completion 2025-09-26 (Estimated)

PRIMARY OUTCOMES:
Respiratory quotient during exercise | Week 1
  Respiratory quotient measured by indirect calorimetry during the low intensity exercise.
Respiratory quotient during exercise | Week 2
  Respiratory quotient measured by indirect calorimetry during the low intensity exercise.
Respiratory quotient during exercise | Week 3
  Respiratory quotient measured by indirect calorimetry during the low intensity exercise.
Respiratory quotient during exercise | Week 4
  Respiratory quotient measured by indirect calorimetry during the low intensity exercise.
Respiratory quotient during exercise | Week 8
  Respiratory quotient measured by indirect calorimetry during the low intensity exercise.
Respiratory quotient during exercise | Week 12
  Respiratory quotient measured by indirect calorimetry during the low intensity exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, AURA, France

IPD SHARING:
Plan to Share IPD: No